CLINICAL TRIAL: NCT00377585
Title: A Phase II/III, Observer-blind, Multi-Country, Multi-Centre, Randomized Study to Demonstrate the Superiority in Terms of Immunogenicity of Adjuvanted Influenza Vaccine Administered in Adults Aged 50 Years and Older Compared to Fluarix™
Brief Title: Demonstrate the Superiority of the Immune Response of Adjuvanted Influenza Vaccine Induced in an Adult Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 104888
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Elderly; Improved vaccine; Influenza; Influenza disease
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

INTERVENTIONS:
Biological: Fluarix
Biological: adjuvanted influenza vaccine
  Other Names: Fluarix

SUMMARY:
The study is designed to demonstrate a meaningful difference in immunogenicity between the candidate adjuvanted vaccine compared to the licensed Fluarix vaccine in subjects aged 50 years and above.

A control group in younger adults aged 18 to 40 years was included.

DETAILED DESCRIPTION:
This is a study to demonstrate the superiority of the immune response of adjuvanted influenza vaccine induced in an adult population.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must be healthy adults 18-40 years or >/= 50 years.

Exclusion Criteria:

* Subjects will be excluded if they take/have taken chronically high doses of immunosuppressants or other immune modifying drugs within six months before vaccination, or immunoglobulins or blood products within three months before vaccination, or any investigational product within 30 days before vaccination, or a licensed vaccine within 2 (inactivated) to 4 (live) weeks before vaccination, if women are pregnant or lactating, or if subjects have acute clinically significant disease or an immunosuppressive/deficient condition, or have contra-indications to influenza vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3350
Dates: Start 2006-09-22; Study Completion 2007-01-30 (Actual)

PRIMARY OUTCOMES:
To demonstrate that the immune response induced by the adjuvanted influenza vaccine in the elderly is superior to that induced by Fluarix, for each vaccine strain

SECONDARY OUTCOMES:
To evaluate in all subjects, the safety, the humoral response and the cell-mediated immune (CMI) response of the adjuvanted influenza vaccine and Fluarix

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (10):
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
- GSK Investigational Site, Ghent, Belgium
- Germany (8):
  - GSK Investigational Site, Messkirch, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Langquaid, Bavaria
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
- Norway (7):
  - GSK Investigational Site, Bekkestua
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Fredrikstad
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Haugesund
  - GSK Investigational Site, Paradis
  - GSK Investigational Site, Skien

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 104888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study104888 are summarised with study 107509 on the GSK Clinical Study Register.
- Available data/document: Study Protocol: 104888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register